CLINICAL TRIAL: NCT01932346
Title: Using Non-invasive Near Infra-red Spectroscopy to Measure the Regional Tissue Perfusion in Patients Receiving Off-pump Coronary Artery Bypass Graft Surgery
Brief Title: Using Near Infra-red Spectroscopy to Measure Tissue Perfusion in Patients Receiving Coronary Artery Bypass Graft Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201201016RIC
Record Dates: First submitted 2013-08-12; First posted 2013-08-30 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Coronary Artery Disease
Keywords: near infra-red spectroscopy, coronary artery bypass grafting
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Near infra-red spectroscopy (NIRS) was used to measure the tissue perfusion of the cerebral cortex with two noninvasive adhesive patches in recent years. This study is designed to compare the regional tissue perfusion of different body areas in patients receiving coronary artery bypass surgery under general anesthesia. The NIRS data will also be used to compare with other routine physiological monitors in the surgery.

DETAILED DESCRIPTION:
Study Design:

Prospective observational study

Target Number of Participants:

To recruit 50 patients into this study.

Patient Selection:

1. Patients scheduled for elective coronary artery bypass surgery.
2. The American Society of Anesthesiologists physical status classification system(ASA) Class I~III
3. Age ≧20 y/o, ≦75 y/o

Exclusion Criteria:

1. ASA Class IV
2. Current skin lesion over the sites where the NIRS patches are designed to be attached.
3. Patients received cardiopulmonary bypass during the surgery.
4. Patients with previous history of allergy to the NIRS patches.

Study Method:

After the induction of anesthesia, four NIRS patches are attached to the patients on the following sites:

1. Biceps brachii muscle area
2. Gastrocnemius muscle area
3. Posterior side of neck
4. central part of the forehead

The four non-invasive NIRS patches are only to measure the tissue oxygen saturation and have no other physiological effects on the participants.

The data will be collected every 5 minutes until the surgery is completed. The data from other routine monitors used during the surgery (including hear rate, blood pressure, and mixed venous saturation) will also be used to compare with the data from NIRS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧20 years old, ≦75 years old
* Patients scheduled for elective coronary artery bypass surgery
* ASA Class I~III

Exclusion Criteria:

* Patients scheduled for cardiopulmonary bypass
* Allergy for NIRS

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective coronary artery bypass surgery and age ≧20 years old, ≦75 years old
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of tissue oxygen saturation (StO2) | every 5 minute, from the induction of anesthesia to the end of the surgery, estimated duration: 4 hours
  The measured tissue oxygen saturation is shown in the form of percentage (0~100%).

CONTACTS AND LOCATIONS:
Overall Officials: Po-Yuan Shih, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Using non-invasive near infra-red spectroscopy to measure the regional tissue perfusion in patients receiving off-pump coronary artery bypass graft surgery, Taipei, Taiwan